CLINICAL TRIAL: NCT01549470
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Multiclade HIV-1 DNA Plasmid Vaccine, VRC-HIVDNA009-00-VP, in Uninfected Adult Volunteers in Uganda
Brief Title: Evaluating the Safety of and Immune Response to an HIV Vaccine in Healthy, HIV-Uninfected Adults in Uganda
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RV 156; 10468 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study vaccine (Experimental): Participants in this arm will receive a total of three doses of study vaccine: the first dose at Day 0, the second dose at Day 28 (plus or minus 7 days), and the third dose at Day 56 (plus or minus 7 days). Each dose will consist of a 1-mL injection (dose strength 4 mg/mL) and will be administered by IM injection in the deltoid muscle.
  Interventions: Biological: VRC-HIVDNA009-00-VP
- Placebo vaccine (Placebo Comparator): Participants in this arm will receive a total of three doses of a placebo vaccine: the first dose at Day 0, the second dose at Day 28 (plus or minus 7 days), and the third dose at Day 56 (plus or minus 7 days). Each dose will consist of a 1-mL injection and will be administered by IM injection in the deltoid muscle.
  Interventions: Biological: Placebo vaccine

INTERVENTIONS:
Biological: VRC-HIVDNA009-00-VP — Administered as a 4 mg/mL dose by IM injection in the deltoid muscle using the Biojector 2000 needle-free injection management system.
  Arms: Study vaccine
Biological: Placebo vaccine — Administered as a 1-mL dose by IM injection in the deltoid muscle using the Biojector 2000 needle-free injection management system.
  Arms: Placebo vaccine

SUMMARY:
Currently, no vaccine prevents HIV infection. This study will test the safety and immune responses of an HIV-1 DNA vaccine in HIV-uninfected adults in a Ugandan population.

DETAILED DESCRIPTION:
The global HIV/AIDS epidemic continues to increase at unacceptably high levels, and there is not yet an effective prevention method for HIV infection. This study will test the safety and immune responses of a preventive HIV vaccine, VRC-HIVDNA009-00-VP, which is a multiclade HIV-1 DNA plasmid vaccine.

This study will seek to enroll 30 participants, randomly assigning 15 participants each to the study vaccine arm and the placebo vaccine arm. Three doses of the vaccine will be given by intramuscular (IM) injection using the Biojector 2000 needle-free injection management system: the first dose at Day 0 (entry), second dose at Day 28 (within 7 days before or after Day 28), and third dose at Day 56 (within 7 days before or after Day 56). Participants will attend two screening visits and visits at Days 0 (entry), 2, 14, 28, 30, 42, 56, 58, 70, 84, 168, 252, and 336. At most visits, participants will give a medical history and undergo a physical exam, blood draw, and urine collection. For women, a pregnancy test will be given at each study injection visit. Participants also will be instructed to maintain a diary of local and systemic reactions for 7 days after each injection. They also will be provided with a ruler to measure erythema, induration, or other observable reactions and a thermometer to record temperature on a daily basis.

ELIGIBILITY:
Inclusion criteria:

* 18 to 40 years old
* Available for follow-up for the duration of the study (13 months)
* Satisfactory completion of an Assessment of Understanding prior to enrollment defined as 90% correct with three opportunities to take test. Errors will be reviewed with volunteer after each test.
* Able and willing to sign the informed consent form
* Willing to receive HIV counseling and testing in accordance with Ugandan Ministry of Health Guidelines
* Willing to discuss HIV infection risks and not currently at high-risk of HIV as defined by responses to a standard questionnaire found in the protocol, agree not to engage in high-risk behavior for HIV during the study as defined by protocol, and amenable to risk-reduction counseling
* Willing to permit a home visit after one of two screening visits
* In good general health without clinically significant medical history
* Physical examination and laboratory results without clinically significant findings within 45 days prior to first injection
* Can understand and read English or Luganda

Within 45 days prior to enrollment, must meet following criteria:

* Hemoglobin greater than 11.0 g/dL for women and 12.5 g/dL for men
* White blood cell (WBC) count: 3,300 to 12,000 cells/mm^3 (in the absence of clinical or pathological etiology)
* Differential either within institutional normal range or accompanied by site physician approval. More information on this criterion can be found in the protocol.
* Total lymphocyte count greater than 800 cells/mm^3 (in the absence of clinical or pathological etiology)
* Platelets = 125,000 to 550,000 cells/mm^3
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) less than 1.25 times the upper limit of normal (ULN)
* Serum creatinine less than ULN
* Normal urinalysis defined as dipstick with negative glucose, negative or trace protein, and negative or trace hemoglobin (blood)
* Negative Food and Drug Administration (FDA)-approved HIV blood test
* Negative serum hepatitis B surface antigen test
* Negative serum hepatitis C antibody test
* Negative urine or serum-human chorionic gonadotropin (HCG) pregnancy test for all women. A female participant must meet one of the following criteria from 21 days prior to vaccination until 3 months following the last vaccination:

  1. No reproductive potential because of a hysterectomy, bilateral oophorectomy, or tubal ligation. Documentation from qualified medical doctor must be obtained for confirmation of procedure, OR
  2. Participant agrees to consistently practice contraception at least 21 days prior to vaccination and throughout the duration of the study by one of the following methods:

     1. condoms, male or female, with or without a spermicide
     2. diaphragm or cervical cap with spermicide
     3. intrauterine device
     4. contraceptive pills, Norplant or Depo-Provera
     5. male partner has previously undergone a vasectomy for which there is documentation
     6. abstinence from sexual activity
* Men should not take part in this study if they plan to father a child between the first vaccination and 3 months after the last vaccination. Men should consistently use a condom, provide documentation of vasectomy from qualified medical doctor, practice abstinence of sexual activity, OR his female partner should use one of the following methods:

  1. female condoms, with or without spermicide
  2. diaphragm or cervical cap with spermicide
  3. intrauterine device
  4. contraceptive pills, Norplant or Depo-Provera

Exclusion Criteria

* Woman who is breast-feeding
* Has received HIV vaccines in a prior clinical trial
* Has received immunosuppressive or cytotoxic medications within the past 6 months with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis
* Has received blood products within 120 days prior to HIV screening
* Has received immunoglobulin within 60 days prior to HIV screening
* Has received live attenuated vaccines within 30 days prior to initial study vaccine administration
* Has received investigational research agents within 30 days prior to initial study vaccine administration
* Has received medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration
* Is receiving current anti-tuberculosis (TB) prophylaxis or therapy
* History of a serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
* History of autoimmune disease or immunodeficiency
* History of asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years or that requires the use of oral or intravenous corticosteroids
* History of diabetes mellitus (type I or II), with the exception of gestational diabetes
* History of thyroid disease including history of thyroidectomy and diagnoses that required medication within the past 12 months
* History of serious angioedema episodes within the previous 3 years or requiring medication in the previous 2 years
* History of hypertension controlled by medication or is more than 140/90 at enrollment
* History of bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
* History of active syphilis documented by exam or serology unless positive serology is due to remote (greater than 6 months) treated infection or positive rapid plasma reagin (RPR)/venereal disease research laboratory (VDRL) is not associated with positive treponemal specific serology
* History of malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study
* History of seizure disorder other than febrile seizures under the age of 2, seizures secondary to alcohol withdrawal more than 3 years ago, or a singular seizure not requiring prolonged treatment more than 3 years ago
* History of asplenia or any condition resulting in the absence or removal of the spleen
* History of psychiatric condition that precludes compliance with the protocol, past or present psychoses, past or present bipolar disorder or suicidal ideation
* History of any medical, psychiatric, or social condition or occupational or other responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence or a volunteer's ability to give informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Local reactogenicity signs and symptoms | Measured through Week 48 visit
Systemic reactogenicity signs and symptoms | Measured through Week 48 visit
Laboratory measures of safety | Measured through Week 48 visit
All adverse experiences and serious adverse experiences | Measured through Week 48 visit
HIV-specific cellular immune responses | Measured through Week 48 visit
  As measured by interferon (IFN)-gamma enzyme-linked immunosorbent spot (ELISpot) and intracellular cytokine assay using frozen peripheral blood mononuclear cells (PBMCs) and overlapping peptide pools representing the immunogens.

SECONDARY OUTCOMES:
Lymphoproliferative responses | Measured through Week 48 visit
Cytotoxic T lymphocyte (CTL) measured by chromium release assays | Measured through Week 48 visit
Antibody immune responses as measured by enzyme-linked immunosorbent assay (ELISA) | Measured through Week 48 visit
Neutralizing antibody assays | Measured through Day 70

CONTACTS AND LOCATIONS:
Overall Officials: Fred Wabwire-Mangen, MB ChB, DTM&H, MPH, PhD, Study Chair — Makerere Univ. Institute of Public Health, Dept. of Epidemiology and Biostatistics
Locations (1):
- Makerere University Walter Reed Project (MUWRP), Kampala, Uganda

REFERENCES:
- [Background] Graham BS. Clinical trials of HIV vaccines. Annu Rev Med. 2002;53:207-21. doi: 10.1146/annurev.med.53.082901.104035. PMID 11818471